CLINICAL TRIAL: NCT06357819
Title: INSTI® HCV (Hepatitis C Virus) Antibody Self-Test Contrived Result Interpretation
Status: Completed | Type: Observational
Sponsor: bioLytical Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: CLS-017A; HSTAR010 (Other: HSTAR Programme); EZIMOM012 (Other: Ezintsha)
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C Self Test; Hepatitis C Rapid Test; HCV antibody; INSTI HCV Self Test
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mock Result Interpretation: Testing with non-functional devices (Mock-ups) that are modified to display contrived results to assess the ability of previously untrained users to correctly interpret one of the possible results as defined by each device manufacturer (e.g., Negative/Non-Reactive, Positive/Reactive, Invalid etc.)
  Interventions: Device: INSTI HCV Self Test

INTERVENTIONS:
Device: INSTI HCV Self Test — Each participant was provided with contrived INSTI membrane units by the study observer, in random order, and was asked to interpret the results using the INSTI HCV ST Instructions for Use.

SUMMARY:
The purpose of this Interpretation Assessment was to document if "lay" people, non-professional and inexperienced in self-testing, were able to successfully perform the steps to use a Hepatitis C Virus (HCV) Self-Test (HCVST) device, without product familiarization [demonstration].

DETAILED DESCRIPTION:
The intent of this study was to collect data regarding the result interpretation of contrived results of INSTI HCV ST. The contrived test devices refers to mock test devices pre-made by bioLytical Laboratories Inc. Each contrived/mock test device was assigned to an ID number to be randomly provided to the participants.

Primary Objectives were to document and record the following:

•Successful interpretation of contrived test results using mock test devices (strong positive, weak positive, negative and a range of invalid results).

Depending on the device being evaluated participants received a contrived INSTI® HCV Antibody Self Test membrane unit.

Participants were asked to interpret "mock" results [read contrived device results using the reference chart in the Instructions for Use (IFU)].

Participants were recruited from the Ezintsha Research Site which was a low-prevalence area and the Yeoville Harm Reduction Site which was a high-prevalence area in the city of Johannesburg in the Republic of South Africa. For the purposes of this assessment, the participant population was the general population. The participants did not have any experience in conducting any rapid diagnostic self-test using standard test kits, nor were they familiar with the prospective HCVST devices prior to entering into this mock result interpretation assessment.

ELIGIBILITY:
Inclusion Criteria:

* Understands and sign the written informed Consent form
* Able to complete the required testing on the allocated testing day[s]
* Able to speak/read English
* ≥18 years of age
* Provide a level of education (minimum grade 7)

Exclusion Criteria:

* Does not meet the inclusion criteria
* A practicing medical healthcare professional [doctor, nurse or counsellor that performs testing with Rapid Tests]
* Has used blood-based RDT for self-testing previously, either HIV or HCV
* Any condition which, in the opinion of the facilitator, would make the participant unsuitable or unsafe for enrolment or could interfere with the completion of the mock result interpretation assessment, consent form and questionnaire etc. or bias the outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were recruited and enrolled from high and low HCV-prevalence areas to participate in mock result interpretation of INSTI HCV Selt Tests.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2023-12-17 (Actual)

PRIMARY OUTCOMES:
Successful Interpretation of contrived devices | 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- bioLytical Laboratories Inc., Richmond, British Columbia, Canada